CLINICAL TRIAL: NCT06267833
Title: The Effect of Adding Trunk and Upper Extremity Exercises to the Otago Exercise Program on Balance Performance, Fall Risk, and Fear of Falling in Older Adults
Brief Title: The Effect of Trunk and Upper Extremity Exercises Added to the Otago Exercise Program
Acronym: Otago Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Gizem Murat, Research Assistant, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MSKUSBFFTR01
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Geriatrics; Balance; Exercise; Fall Prevention
Keywords: Geriatrics; Balance; Fall prevention; Mobil game; telerehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Receiving the Otago exercise program
  Interventions: Behavioral: exercise
- Study group 1 (Experimental): Receiving additional trunk and upper extremity exercises with traditional methods added to the Otago exercise program
  Interventions: Behavioral: exercise
- Study group 2 (Experimental): Receiving additional trunk and upper extremity exercises with mobile game method added to the Otago exercise program
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — In the exercise protocol, a personalized, home-based, 30-minute Otago exercise program consisting of strength, balance, and walking exercises performed three times a week will be implemented for 8 weeks with home visits and telerehabilitation sessions (via Videoconferencing) under the supervision of the responsible researcher. In addition to the Otago exercise program, trunk and upper extremity exercises (totaling 45 minutes) will be implemented in study group 1 using traditional methods and in study group 2 using the mobile game method.

SUMMARY:
This study is designed to investigate the effect of adding trunk and upper extremity exercises in traditional and mobile game formats to the Otago exercise program on balance performance, fall risk, and fear in older adults. A randomized controlled, cross-sectional, single-blind (evaluator) study will be conducted with 36 older adults aged 65 and older enrolled at Muğla Sıtkı Koçman University (MSKÜ) Elderly Studies Application and Research Center. Participants will be divided into three randomized groups: control group (12 individuals receiving the Otago exercise program), study group 1 (12 individuals receiving additional trunk and upper extremity exercises with traditional methods added to the Otago exercise program), and study group 2 (12 individuals receiving additional trunk and upper extremity exercises with mobile game method added to the Otago exercise program). Participant demographics informations will be recorded in Form 1. Participants' cognitive functions , levels of independence in activities of daily living, fall risk , and fear of falling will be evaluated. Balance performance will be assessed using the Mini Balance Evaluation Systems Test (Mini-BESTest), portable computerized kinetic balance measurement (SportKAT 650-TS), "5 Times Sit-to-Stand" and "Four-Stage Balance Test" from the Otago Exercise Program. Participants' body sway will be assessed simultaneously with the second part of the Mini-BESTest using a mobile application. All assessments will be conducted by a researcher blinded to the exercises, both before and after the exercises, in a one-on-one face-to-face setting. In the exercise protocol, a personalized, home-based, 30-minute Otago exercise program consisting of strength, balance, and walking exercises performed three times a week will be implemented for 8 weeks with home visits and telerehabilitation sessions (via Videoconferencing) under the supervision of the responsible researcher. In addition to the Otago exercise program, trunk and upper extremity exercises (totaling 45 minutes) will be implemented in study group 1 using traditional methods and in study group 2 using the mobile game method. Telerehabilitation sessions will be conducted via an Android-based tablet if the study is supported by Tübitak 1002 A Rapid Support Module. Individual smartphones of participants will be used if the study is not supported. All questionnaires, scales, and tests used in the initial assessments will be repeated at the end of the 8-week exercise protocol for all participants.

ELIGIBILITY:
Inclusion Criteria:

* To be aged 65 years and older.
* To have the ability to speak, read, comprehend, and write in Turkish.
* To have a body mass index <35 kg/m2 (not being severely or morbidly obese).
* To have experienced one or more falls within the past 1 year.
* To possess cognitive abilities enabling the understanding and implementation of the educational sessions to be conducted in the study (having scored ≥ 24 points on the Mini-Mental State Examination).
* To be able to perform daily activities independently (scoring 5-6 points on the Katz Activities of Daily Living Scale).
* To demonstrate a reach performance of ≥ 16 centimeters in the Functional Reach Test.
* To be able to walk independently (regardless of the use of walking aids).
* To have internet connectivity at home.
* To permit the implementation of exercise protocols under the supervision of the researcher in the home environment.
* To allow for periodic home visits by the researcher for the implementation of exercise protocols.
* To agree to have a physically suitable area in the home for exercise protocols or to make necessary arrangements to render the home environment suitable for exercise.

Exclusion Criteria:

* To have absolute contraindications for strength and aerobic exercises.
* To have chronic pain in the lower body and extremities.
* To have a disorder related to the vestibular system.
* To engage in regular exercise that may affect performance outcomes.
* To decline participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mini BESTest | 15 minutes
  Mini Balance Evaluation Systems Test

SECONDARY OUTCOMES:
Functional Reach Test | 3 minutes
  Assessment risk of falling
International Falls Efficacy Scale | 10 minutes
  Assessment fear of falling

IPD SHARING:
Plan to Share IPD: No